CLINICAL TRIAL: NCT00789685
Title: A Phase I/II Open-Label Study to Assess the Safety, Tolerability and Preliminary Efficacy of FP-1201 (Recombinant Human Interferon Beta) in the Treatment of Patients With Acute Lung Injury and Acute Respiratory Distress Syndrome.
Brief Title: Safety, Tolerability and Preliminary Efficacy of FP-1201 in ALI and ARDS. Phase I/II
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Faron Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FPCLI001
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Open label
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome | interventions — Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon Beta (Experimental): Interferon Beta
  Interventions: Drug: Interferon Beta

INTERVENTIONS:
Drug: Interferon Beta — Interferon Beta administered intravenously daily for 6 days. Doses of 0.12 MIU, 1.2 MIU, 2.7 MIU or 6.0 MIU (dose escalation phase) or 2.7 MIU (dose expansion phase) were administered.
  Other Names: FP-1201; IFN-beta

SUMMARY:
The purpose of this study was to assess the safety, tolerability and preliminary efficacy of FP-1201 (Interferon Beta) in patients with Acute Lung Injury (ALI) and Acute Respiratory Distress Syndrome (ARDS).

DETAILED DESCRIPTION:
This was a phase I/II open-label study to assess the safety, tolerability and preliminary efficacy of FP-1201 (IFN β-1a) in the treatment of patients with ALI and ARDS.

The primary objective in the study was to evaluate the safety and tolerability of FP-1201 in patients with ALI/ARDS and to assess the safety, tolerability and preliminary efficacy of the optimum tolerated dose (OTD) in patients likely to derive clinical benefit.

The study consisted of a dose escalation phase to determine the maximum tolerated dose (MTD) and OTD followed by a separate cohort expansion phase in which the OTD was administered.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients with ALI/ARDS confirmed by the combination of the following diagnostic criteria:

  * An initiating clinical condition (e.g. sepsis, pneumonia, aspiration pneumonia, pancreatitis etc.)
  * Acute onset
  * Bilateral infiltrates documented by chest radiograph at end-aspiratory position
  * The absence of clinical evidence of left atrial hypertension
  * ALI: partial pressure of oxygen (PaO2) / fraction of inspired oxygen (FiO2) ratio ≤300 mmHg in a stable state after the patient has adapted to standardised ventilation. (Within the UK this equates to <40kPa)
  * ARDS: PaO2 /FiO2 ≤200 mmHg in a stable state after the patient has adapted to standardised ventilation. (Within the UK this equates to <26.7kPa)
* Provision of signed written informed consent from the patient or patients legally authorized representative.
* Age greater than or equal to 18.
* Initiation of study drug within 48 hours of the diagnosis of ALI/ARDS.
* All patients at entry are required to be receiving mechanical ventilatory support.
* Only patients who are considered suitable for active life support should be enrolled in the study.
* No clinical evidence of left atrial hypertension that would explain the pulmonary infiltrates; if measured the pulmonary arterial wedge pressure should be less than or equal to 18mmHg

Exclusion Criteria:

* Patients with burns.
* Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.
* Patients with significant Chronic Obstructive Pulmonary Disease requiring ongoing treatment e.g. chronic use of oxygen or ventilatory support at home prior to admission.
* Patients with primary lung cancer or the presence of secondary metastases in the lungs.
* Patients requiring treatment for congestive heart failure.
* Patients receiving renal dialysis therapy for chronic renal failure.
* Patients taking immunomodulatory therapy or oral steroids on admission.
* Prior use of interferon.
* Inability to maintain blood pressure to ensure adequate end organ perfusion. It should be noted that the use of plasma colloids or vasopressor agents is allowed to achieve the maintenance of blood pressure.
* Current participation in another experimental treatment protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Bellingan, MD, Principal Investigator — University College London Hospital; Martin Kuper, MD, Principal Investigator — Whittington Hospital; Martin Stotz, MD, Principal Investigator — St Mary's Hospital, London; Richard Beale, MD, Principal Investigator — St Thomas' Hospital; Mathew Wise, MD, Principal Investigator — University Hospital of Wales; Alexander Binning, MD, Principal Investigator — Western Infirmary; Alan Davidson, MD, Principal Investigator — Victoria Infirmary; Timothy Walsh, MD, Principal Investigator — Edinburgh Royal Infirmary
Locations (8):
- United Kingdom (8):
  - University Hospital of Wales, Cardiff
  - Edinburgh Royal Infirmary, Edinburgh
  - Western Infirmary, Glasgow
  - Victoria Infirmary, Glasgow
  - Whittington Hospital, London
  - University College London Hospital, London
  - St Thomas' Hospital, London
  - St Mary's Hospital, London

REFERENCES:
- [Background] Kiss J, Yegutkin GG, Koskinen K, Savunen T, Jalkanen S, Salmi M. IFN-beta protects from vascular leakage via up-regulation of CD73. Eur J Immunol. 2007 Dec;37(12):3334-8. doi: 10.1002/eji.200737793. PMID 18034430
- [Result] Bellingan G, Maksimow M, Howell DC, Stotz M, Beale R, Beatty M, Walsh T, Binning A, Davidson A, Kuper M, Shah S, Cooper J, Waris M, Yegutkin GG, Jalkanen J, Salmi M, Piippo I, Jalkanen M, Montgomery H, Jalkanen S. The effect of intravenous interferon-beta-1a (FP-1201) on lung CD73 expression and on acute respiratory distress syndrome mortality: an open-label study. Lancet Respir Med. 2014 Feb;2(2):98-107. doi: 10.1016/S2213-2600(13)70259-5. Epub 2013 Dec 23. PMID 24503265
- See also: Sponsor's website — http://www.faronpharmaceuticals.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Interferon Beta
Started | 37
Completed | 25 (Completed the study to Day 28)
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: The safety population was used for summaries of demographic and other baseline characteristics
Groups:
- Safety Population: Safety population includes all patients who received at least one dose of study medication, and was used for summaries of demographic and other baseline characteristics
Arm/Group | Safety Population
Number analyzed (Participants) | 37
Age, Continuous [Mean (Full Range); unit: years] | 52.6 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 31
  Black or African | 3
  South American | 1
  Asian | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 37

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Treatment Emergent Events
Description: Treatment-emergent adverse events (TEAEs) in safety population
Time Frame: From first dose up until Day 28
Population: Patients included in Safety population
Measure: Number; unit: Number of patients
Groups:
- Safety Population: Safety population includes all patients who received at least one dose of study medication
Arm/Group | Safety Population
Number analyzed (Participants) | 37
Number of patients
  TEAEs | 37
  Severe TEAEs | 30
  Serious TEAEs | 22
  Drug-Related TEAEs | 20
  Serious Drug-Related TEAEs | 8
  TEAEs leading to withdrawal | 6

2. Primary Outcome: All Cause Mortality at Day 28
Description: The primary efficacy variable was all cause mortality at Day 28 following commencement of treatment
Time Frame: 28 days following commencement of therapy
Population: Patients included in Safety population
Measure: Number; unit: percentage of patients who died
Arm/Group | Safety Population
Number analyzed (Participants) | 37
percentage of patients who died | 8.1

3. Secondary Outcome: All Cause Mortality Rate at 6 Months
Description: A long-term secondary efficacy variable was all cause mortality at 6 months following commencement of treatment
Time Frame: 6 months following commencement of therapy
Population: Number of patients whose survival status at 6 months was known
Measure: Number; unit: percentage of patients who died
Arm/Group | Safety Population
Number analyzed (Participants) | 36
percentage of patients who died | 11.1

ADVERSE EVENTS:
Time Frame: Over the course of the study (Days 1 - 28) and at withdrawal
Description: Adverse Events (AEs) were reviewed and documented from the time the first dose was given up until Day 28. AEs were also reviewed and documented at the withdrawal visit.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 22/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=37)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) — Fatal outcome
Cardiac Arrest (Cardiac disorders) | 2 (4)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Sinus Tachycardia (Cardiac disorders) | 1 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoglobin Decreased (Investigations) | 2 (2)
Klebsiella Sepsis (Infections and infestations) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Clostridial Infection (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 2 (2) — Fatal outcome
Septic Shock (Infections and infestations) | 1 (1) — Fatal outcome
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1)
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=37)
Haemoglobin Decreased (Investigations) | 12 (22)
Electrocardiogram T Wave Inversion (Investigations) | 2 (2)
Nasogastric Output High (Investigations) | 2 (2)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1)
Blood Sodium Increased (Investigations) | 1 (1)
Electrocardiogram QT Prolonged (Investigations) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 1 (1)
Troponin T Increased (Investigations) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 9 (35)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (11)
Constipation (Gastrointestinal disorders) | 9 (10)
Mouth Ulceration (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Faecal volume increased (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Candidiasis (Infections and infestations) | 4 (5)
Clostridial Infection (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Oral Candidiasis (Infections and infestations) | 2 (2)
Staphylococcal Infection (Infections and infestations) | 1 (2)
Abdominal Sepsis (Infections and infestations) | 1 (1)
Bacterial Infection (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 1 (1)
Escherichia Infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Klebsiella Infection (Infections and infestations) | 1 (1)
Lung Infection Pseudomonal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia Cytomegaloviral (Infections and infestations) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1)
Urinary Tract Infection Fungal (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 10 (11)
Agitation (Psychiatric disorders) | 5 (6)
Confusional State (Psychiatric disorders) | 4 (5)
Delirium (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 (1)
Pyrexia (General disorders) | 11 (17)
Hyperpyrexia (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Generalised Oedema (General disorders) | 1 (1)
Influenza Like Illness (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (8)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Arrhythmia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Right Ventricular Hypertrophy (Cardiac disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (6)
Oedema Peripheral (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Cavitation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Gas Exchange Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (6)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (7)
Haemorrhage (Vascular disorders) | 2 (2)
Post Procedural Haemorrhage (Vascular disorders) | 2 (2)
Cerebral Infarction (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Extremity Necrosis (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 4 (6)
Polyuria (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Renal Pain (Renal and urinary disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1)
Peroneal Nerve Palsy (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Collapse of Lung (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous Emphysema (Injury, poisoning and procedural complications) | 1 (1)
Genital Swelling (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Penile Oedema (Reproductive system and breast disorders) | 1 (1)
Scrotal Oedema (Reproductive system and breast disorders) | 1 (1)
Scrotal Swelling (Reproductive system and breast disorders) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 1 (3)
Critical Illness Polyneuropathy (Musculoskeletal and connective tissue disorders) | 2 (2)
Rib Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Herpes Simplex Ophthalmic (Eye disorders) | 1 (1)
Vitreous Floaters (Eye disorders) | 1 (1)
Deafness Unilateral (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Review by sponsor of related publication & communications